CLINICAL TRIAL: NCT05488704
Title: The Effect of Nonstress Test Device Noise Level on Stress Parameters in Primiparous Pregnant Women
Status: Active, not recruiting | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Other Study IDs: 35620
Record Dates: First submitted 2022-07-26; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Stress; Noise Exposure; Prenatal Stress; Prenatal Care Late; Pregnancy Related
Keywords: Adrenocorticotropic Hormone; Pregnancy; Noise; Prenatal Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Cortisol and Saliva ACTH samples were taken to measure the stress levels of pregnant women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CONTROL GROUP: Control Group [NST device volume turned off]
  Interventions: Diagnostic Test: Stress Parameters Measurement
- Intervention Group I: Intervention Group I [NST device volume 1-35 dB(A)]
  Interventions: Diagnostic Test: Stress Parameters Measurement
- Intervention Group II: Intervention Group II [NST device volume 36-60 dB(A)]
  Interventions: Diagnostic Test: Stress Parameters Measurement
- Intervention Group III: Intervention Group III [61 dB( A) and above]
  Interventions: Diagnostic Test: Stress Parameters Measurement

INTERVENTIONS:
Diagnostic Test: Stress Parameters Measurement — Pre-Test (0-2 minutes before NST starts) - Measurement of vital parameters (Pre-Test)
  * Glucose measurement
  * Taking Salivary Cortisol and Saliva ACTH samples
  * Filling the Spielberger State Anxiety Inventory
    • Starting NST by controlling the noise level Interim Test-(NST 10th minute) - Measurement of vital parameters (Intermediate Test)
  * Taking Salivary Cortisol and Saliva ACTH samples
  * Filling the Spielberger State Anxiety Inventory
    • Termination of NST after 20 minutes Final Test(within 0-2 minutes after NST is over)
  * Measurement of vital parameters
  * Glucose measurement
  * Taking Salivary Cortisol and Saliva ACTH samples
  * Filling the Spielberger State Anxiety Inventory After Data Collection - Recording of data
  * Centrifugation and analysis of saliva samples taken

SUMMARY:
Introduction: Prenatal tests can increase the stress levels of pregnant women. One of the tests performed to evaluate fetal health during pregnancy is the Nonstress Test (NST).

Objective: To evaluate the effect of NST device noise level on stress parameters in primiparous pregnant women.

Method: A randomized controlled, prospective study was conducted with 44 pregnant women in a State Hospital in Istanbul/Turkey between 01.02.2021 and 01.10.2021.

Personal Information Form, Spielberger State Anxiety Inventory, Hillrom Welch Allyn Connex Spot Monitor, Gluco Dr Glucometer, Extech SL 400 Personal Noise Dosimeter, Sennheiser HD 450BT ANC Over-Ear Bluetooth Headset, Eppendorf Tube, Philips Avalon FM20 NST were used to collect data. A p value of <.05 was considered significant in the statistical evaluation.

DETAILED DESCRIPTION:
A number of tests are used to evaluate fetal health during pregnancy. One of these tests is the NST. NST is a frequently used fetal evaluation method in gynecology clinics/services during pregnancy and labor. The sound levels of the NST device are created in a way that the healthcare professional can adjust, and at the same time, the average dB(A) range of the sound levels is not known. It has been stated in many studies that noise causes stress in individuals, and that the stress experienced in pregnant women is associated with negative maternal and neonatal outcomes. It is important to evaluate NST noise levels and stress parameters in order to maintain NST, which is a frequently used fetal evaluation method in the prenatal period in clinical practice, without causing maternal stress and to prevent possible negative consequences. With the information to be obtained in line with the results of the research, it is aimed to maintain the noise level of the NST device used by the midwives in the most appropriate sound range for the pregnant women and thus to ensure that the stress levels of the pregnant women are at the lowest level during the procedure.

This study was carried out to evaluate the effect of NST device noise level on stress parameters in primiparous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research,
* Over 18 years old,
* Literate,
* Fluent in Turkish
* 32-42 of your pregnancy. in the week,
* Having a healthy pregnancy,
* No adrenal insufficiency,
* No problems with hearing,
* No psychiatric diagnosis during or before pregnancy,
* No history of infertility,
* Coming to routine pregnancy and NST control,
* Have not had any food or drink for at least two hours before the procedure,
* Primiparous pregnant women without contractions were included.

Exclusion Criteria:

* Pregnant women whose contractions are detected during the NST procedure,
* Pregnant women with deceleration detected in the NST procedure were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Only pregnant women were included in the study.
Study Population: It was decided to make the minimum sample size required in the study by power analysis, taking into account the differences of the pre-test and post-test variables, which are the primary results. More than 2 groups analysis (ANOVA) test in repeated measurements in the calculation, effect size: 0.25, type 1 error rate (α)=0.05, power of the study (1- β) was 0.80 (Type II error= 0.20). Accordingly, the minimum number of samples to be reached was calculated as 40 in total, and the study was completed with 44 samples, taking into account the 10% risk of loss.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2028-07-28 (Estimated)

PRIMARY OUTCOMES:
Does increasing the noise level of the NST device affect If salivary cortisol levels | 01.02.2021-01.10.2021
  Data collection tool used to reach this outcome: Saliva cortisol was measured by a microplate reader with commercially available kit based on ELISA.
Does increasing the noise level of the NST device affect If salivary ACTH levels | 01.02.2021-01.10.2021
  Data collection tool used to reach this outcome: Saliva ACTH was measured by a microplate reader with commercially available kit based on ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Turan, PhD, Study Director — Lecturer
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Aysenur T, Nuran G, Cihan K, Huri B. The Effect of Nonstress Device Noise Level on Stress Parameters in Primigravid Women: A Randomized Controlled Trial. J Midwifery Womens Health. 2024 Mar-Apr;69(2):279-286. doi: 10.1111/jmwh.13581. Epub 2024 Jan 4. PMID 38178318